CLINICAL TRIAL: NCT00567970
Title: A Phase I Dose Finding Pilot Study of Stereotactic Body Radiotherapy for the Treatment of Liver Metastasis
Brief Title: Stereotactic Radiation Therapy in Treating Patients With Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000579232; P30CA015083 (NIH); MC0642 (Other: Mayo Clinic Cancer Center); 06-004336 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Cancer
Keywords: liver metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: quality-of-life assessment
Radiation: stereotactic body radiation therapy

SUMMARY:
RATIONALE: Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase I trial is studying the side effects and best dose of stereotactic radiation therapy in treating patients with liver metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify the maximum tolerated dose of stereotactic radiation therapy in patients with hepatic metastases.
* To determine the toxicity and adverse events profile of this patient population.
* To examine patient response, treatment effect on blood chemistry, and hematology values and patient quality-of-life in this patient population.

OUTLINE: Patients are stratified according to stereotactic radiotherapy level (1 vs 2 vs 3) and the number of liver lesions present (1-2 vs 3-5 vs > 5).

Patients undergo percutaneous placement of metallic fiducial markers within the liver for stereotactic targeting and planning. Patients then undergo 1 fraction of stereotactic radiotherapy within 1 week of the marker placement.

Patients complete Brief Pain Inventory and Brief Fatigue Inventory questionnaires to assess quality of life at weeks 2, 4, 6, 8 and months 3, 6, and 9 after completion of study treatment.

After completion of study treatment, patients are followed for at least 8 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Metastatic liver lesion ≤ 5 cm in dimension
* Willing and able to undergo percutaneous placement of localization seeds

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* Platelet count ≥ 75,000/µL
* Hemoglobin ≥ 9 g/dL
* ANC ≥ 1,500/mL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* AST ≤ 3 x ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to complete questionnaires alone or with assistance
* No medical, social, or economic circumstance, that is likely to prevent adherence with the protocol

PRIOR CONCURRENT THERAPY:

* No prior radiation therapy to the liver
* No chemotherapy ≤ 4 weeks prior to registration
* Able to safely go without chemotherapy for 4 weeks after stereotactic radiotherapy (e.g., patients must not have or need chemotherapy in the 8 weeks [4 weeks prior to and 4 weeks after registration] surrounding stereotactic radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-04-02 (Actual); Primary Completion 2009-02-02 (Actual); Study Completion 2016-04-21 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose

SECONDARY OUTCOMES:
Toxicity profile
Adverse events profile
Quality of life as measured by the Brief Pain Inventory and Brief Fatigue Inventory
Response profile
Physical exam results

CONTACTS AND LOCATIONS:
Overall Officials: Laura A. Vallow, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic - Jacksonville, Jacksonville, Florida, United States